CLINICAL TRIAL: NCT06037304
Title: Quality of Life After Shouldice Repair
Acronym: QoL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shouldice Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: QoL
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Hernia, Inguinal
Keywords: Quality of life; shouldice repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This research project aims to assess the quality of life (QOL) and pain/discomfort experienced by patients who have undergone primary inguinal hernia repair at Shouldice Hospital. Historically, postoperative mortality and symptom improvement have been the main outcomes assessed after hernia surgery, neglecting the patient experience. As QOL gains significance in hernia patient care, this study focuses on evaluating patient QOL before and after surgery, contributing to a better understanding of hernia surgery outcomes.

Study Objectives:

Determine preoperative quality of life. Determine patient-reported quality of life at 1 week after surgery. Determine patient-reported quality of life at 1 month after surgery. Determine patient-reported quality of life at 6 months after surgery. Evaluate changes in quality of life from the preoperative time to 6 months after surgery.

Hypotheses/Research Questions:

Does quality of life change after hernia surgery? What is the quality of life before and after primary unilateral inguinal hernia repair? Does hernia repair improve patient quality of life?

Study Design:

This is a prospective cohort pilot study involving primary unilateral inguinal hernia patients who received Shouldice repair at Shouldice Hospital. It includes chart reviews (medical histories and operative notes) and surveys at preoperative, 1-week, 1-month, and 6-month postoperative time points. Surveys are conducted using the EQ5D3L tool to measure health-related quality of life.

Study Population:

The study population includes male and female patients aged 16-90, of all nationalities and races, capable of English communication, in good general health, who had primary unilateral inguinal hernia repair at Shouldice Hospital. Exclusions encompass patients who had mesh repair, non-inguinal hernias, concurrent hernias, bilateral hernia repair, or emergency surgeries.

Data Collection:

Data is collected from patient survey responses, medical records, and charts. Surveys are administered via email at specific time points. A deferred consent process is used, and participants are informed about their rights and the ability to withdraw. Data is deidentified for privacy.

Duration of Study:

The study is expected to take 14 months, with a 3-month recruitment phase, a 6-month follow-up period, and 5 months for data analysis and write-up. The estimated participation time for each participant is 13 minutes, and no reminders are sent.

Risks and Benefits:

There are no known risks to participants, and no direct benefits are provided. Personal data is protected, and participation is voluntary.

This study aims to contribute valuable insights into the quality of life of hernia surgery patients, particularly those who have undergone open tissue hernia repair at Shouldice Hospital.

DETAILED DESCRIPTION:
The proposed project is a pilot study designed in a prospective cohort manner, on primary unilateral inguinal hernia patients who had a Shouldice repair at the Shouldice Hospital. It includes prospective chart review (medical histories and operative notes) and a qualitative component (surveys). Patients will be emailed 5-7 days before surgery, with information inviting them to participate or read more about this research project, and a link to a full consent form. If patients consent they will be taken directly to the first (preoperative) survey and the same methodology will be used again at 1 week, 1 month, and 6 months after surgery. Contact is made by email using the hospital's current survey site: Simple Survey.

The survey is made up of the EQ5D3L, which is a standardized measurement of QOL (health related). The EQ5D3L contains two parts, one that measures health status through rating 5 questions in terms of having no, some or extreme problems with mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

The second part contains a visual analogue scale called EQVAS where participants rate their overall health from 0- worst imaginable to 100- best imaginable. The choice to use the EQ5D3L was made because it is a commonly used tool, has shown comparable results to other validated surveys like the CCS [6], and the EQ5D3L is a single short way to measure QOL. Although many studies use multiple surveys to assess QOL, for simplicity sake, and to reduce time burden on patients as well as prevent any reduced response rate just the EQ5D3L will be used.

The study population will focus on male and female patients aged 16-90 years of age, standard age of patients accepted for surgery at Shouldice Hospital, who had a Shouldice repair of a primary unilateral inguinal hernia at Shouldice Hospital, all nationalities and races, capable of speaking and reading English, in good general health, and there is no geographic location constraint. As there are no translators nor non-English survey options provided, participants who cannot complete the survey in English are excluded. Patients will be excluded if they underwent a mesh repair, a hernia that was not an inguinal type, a concurrent hernia, bilateral hernia repair, and surgery was deemed an emergency.

We aim to contact 1000 2400 patients to analyze a total of 400 participants. This is based off information gathered by the researchers from the first six weeks of recruitment for this project. this institution from previously done prospective projects. When consent forms were emailed, there was a response rate of 4530%, with a retention of patients meeting the criteria and being sent the follow up surveys at 18%. No dropout rate has been measured/considered as we will gather data for this pilot project to go on with a sample size calculation in the future. The 400 patients were concluded based off a multicenter study that used the EQ5D3L and had similar objectives as this present study. The 2018 study looked at survey responses after Lichtenstein repair with two difference meshes and had sample sizes of 411 and 397. Thus, analyzing 400 patients would allow for a meaningful comparison to open inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

The study population will focus on male and female patients aged 16-90 years of age, standard age of patients accepted for surgery at Shouldice Hospital, who had a Shouldice repair of a primary unilateral inguinal hernia at Shouldice Hospital, all nationalities and races, capable of speaking and reading English, in good general health, and there is no geographic location constraint. As there are no translators nor non-English survey options provided, participants who cannot complete the survey in English are excluded.

Exclusion Criteria:

Patients will be excluded if they underwent a mesh repair, a hernia that was not an inguinal type, a concurrent hernia, bilateral hernia repair, and surgery was deemed an emergency.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study focuses on patients aged 16-90 years who underwent a primary unilateral inguinal hernia repair at Shouldice Hospital. The inclusion criteria encompass both male and female patients of all nationalities and races, capable of communicating in English, in good general health, and who did not undergo emergency surgery. Patients who had mesh repair, hernias other than inguinal, concurrent hernias, bilateral hernia repairs, and those who couldn't complete surveys in English are excluded. The goal is to contact 2,400 patients to ultimately analyze 400 participants, based on recruitment data. Consent forms yielded a 45-30% response rate, with an 18% follow-up survey retention rate. No dropout rate has been measured yet. The choice of 400 patients is based on a similar study that analyzed sample sizes of 411 and 397 in a multicenter study involving Lichtenstein repair with different meshes for meaningful comparison to open inguinal hernia repair.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
EQ5D3L one week after surgery | one week after surgery

SECONDARY OUTCOMES:
EQ5D3L one month after surgery | one month after surgery
EQ5D3L six months after surgery | ix months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Christoph Paasch, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No